CLINICAL TRIAL: NCT00004268
Title: Phase II Study of Midodrine for Neurogenic Orthostatic Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Roberts Pharmaceutical (Industry)
Purpose: Treatment
Other Study IDs: 199/11645; RLI-5894009
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Orthostatic Hypotension
Keywords: cardiovascular and respiratory diseases; disease-related problem/condition; orthostatic hypotension; quality of life; rare disease
MeSH Terms: conditions — Hypotension, Orthostatic; Respiratory Tract Diseases; Rare Diseases | interventions — Midodrine

INTERVENTIONS:
Drug: midodrine

SUMMARY:
OBJECTIVES: I. Study further the safety and efficacy of the alpha-receptor agonist midodrine in patients with neurogenic orthostatic hypotension.

II. Assess the quality of life in these patients with this treatment regimen.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a partially randomized, multicenter study. Patients receive oral midodrine three times a day during weeks 1 and 3-5, then either oral midodrine or placebo for weeks 6-8.

Quality of life is assessed at weeks 3, 6, and 8.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Orthostatic hypotension due to autonomic nervous system failure, i.e.: Fall in systolic blood pressure (supine to standing) of at least 15 mm Hg AND Symptoms of dizziness, lightheadedness, unsteadiness with a severity of 4.5 or less on a 10 point scale in 2 of 3 evaluations over a 3 day period --Prior/Concurrent Therapy-- No concurrent sympathomimetics or alpha-receptor agonists or antagonists No concurrent drug with significant smooth muscle relaxant or constrictive properties e.g., calcium channel blockers At least 30 days since other prior investigational agents --Patient Characteristics-- Hepatic: No coagulopathy Renal: No acute nephritis or chronic renal failure Cardiovascular: No sustained supine hypertension greater than 180/110 mm Hg No congestive heart failure No myocardial infarction within the last 6 months No uncontrolled arrhythmia (ventricular tachycardia or second or third degree heart block not treated with pacemaker) No unstable angina pectoris No history of cerebral vascular accident Other: No pheochromocytoma No thyrotoxicosis No seizure disorder Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, Study Chair — Roberts Pharmaceutical
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States